CLINICAL TRIAL: NCT02310308
Title: Effect of a Sugar-free Chewing Gum Containing Magnolia Bark Extract on the Development of Caries Lesions in Healthy Adult Volunteers: a Randomized Controlled Intervention Trial
Brief Title: Effect of a Sugar-Free Chewing Gum Containing Magnolia Bark Extract on Caries Lesions in Healthy Adult Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor in Community Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1083/L
Record Dates: First submitted 2014-11-24; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Dental Caries
Keywords: Xylitol; Magnolia; chewing gum
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- xylitol chewing gum (Active Comparator): Intervention chewing gum administration Each subject will be instructed to chew 1 or 2 pellets for 5 min 3 times a day (2 in the morning, 2 after the midday meal and 1 in the afternoon). Thus, the total daily intake of magnolol and honokiol in MX group will be 11.9 mg/day. The daily use of the two different chewing gums will be carried out for 12 months.
  Interventions: Dietary Supplement: Chewing gum administration
- Xylitol-magnolia chewing gum (Experimental): Intervention chewing gum administration Each subject will be instructed to chew 1 or 2 pellets for 5 min 3 times a day (2 in the morning, 2 after the midday meal and 1 in the afternoon). Thus, the total daily intake of magnolol and honokiol in MX group will be 11.9 mg/day. The daily use of the two different chewing gums will be carried out for 12 months.
  Interventions: Dietary Supplement: Chewing gum administration
- Control chewing gum (Placebo Comparator): Intervention chewing gum Each subject will be instructed to chew 1 or 2 pellets for 5 min 3 times a day (2 in the morning, 2 after the midday meal and 1 in the afternoon). Thus, the total daily intake of magnolol and honokiol in MX group will be 11.9 mg/day. The daily use of the two different chewing gums will be carried out for 12 months.
  Interventions: Dietary Supplement: Chewing gum administration

INTERVENTIONS:
Dietary Supplement: Chewing gum administration — Intervention chewing gum Each subject will be instructed to chew 1 or 2 pellets for 5 min 3 times a day (2 in the morning, 2 after the midday meal and 1 in the afternoon). Thus, the total daily intake of magnolol and honokiol in MX group will be 11.9 mg/day. The daily use of the two different chewing gums will be carried out for 12 months.

SUMMARY:
The effect of chewing gums containing MBE and xylitol on different variables related to caries and gingivitis in a sample of adult volunteers with a high risk for caries will be evaluated. The main result of that double-blind randomized controlled interventional trial will be that chewing gum containing MBE was more effective in reducing plaque acidogenicity, salivary mutans streptococci concentration and gingival bleeding compared to a xylitol and sugar-free chewing gum.

DETAILED DESCRIPTION:
Introduction

Dental caries incidence in adults is similar to that in children and adolescents, but few caries preventive agents have been evaluated for effectiveness in adult populations. Magnolia bark extract (MBE) is a plant extract obtained from the bark of magnolia that has been widely used in traditional Chinese medicine for 2,000 years, Magnolia officinalis has been used for the treatment of acute pain, diarrhea, coughs and urinary problems. The two main constituents of the bark of this medicinal plant are magnolol and honokiol. They are known to possess a variety of pharmacological properties, including therapeutic-related activities central nervous system inhibition anti-inflammatory effects, antimicrobial activity, antioxidative activity and freeradical scavenging activity. Magnolol andhonokiol have also been reported to inhibit the growth of Streptococcus mutans, Streptococcus sobrinus, Porphyromonas gingivalis, Fusobacterium nucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga gingivalis and Veillonella disper in vitro and reduce the dental caries values in rats. Consequently, the antimicrobial properties of MBE against cariogenic and plaque bacteria have showed promising results. The effect of chewing gums containing MBE and xylitol on different variables related to caries and gingivitis in a sample of adult volunteers with a high risk for caries will be evaluated. The main result of that double-blind randomized controlled interventional trial will be that chewing gum containing MBE was more effective in reducing plaque acidogenicity, salivary mutans streptococci concentration and gingival bleeding compared to a xylitol and sugar-free chewing gum.

Materials and Methods A two-year, placebo-controlled, double-blind, randomized clinical trial sponsored by Perfetti Van Melle that tests the effects on caries lesions development of daily use of a chewing gum containing Magnolia Bark Extract and xylitol will be conducted.

The trial will take place in the dental clinics located in the dental schools of the University of Sassari and Milan. The study will be approved by the Ethical Committee of the University of Sassari.

Study Population Principal inclusion criteria will be age range (30-55 years) and the presence of at least one cavitated caries lesion, but no more than three. Subjects with systemic disease that interfered with the oral ecosystem will be excluded. The caries criterion will be designed to include participants who are at risk of forming new lesions. Sample size for preliminary screening will be calculated on the basis of previous studies regarding caries prevalence (about 26%) in adults [Campus et al, 2011] and relative odds ratio 2.88 of incidence, as reported in literature [Ito et al, 2011]. Thus, the theoretical sample size for preliminary screening will be set to 1200 subjects.

In order to get statistical comparison results, the number of subjects per group to be included in the analysis will be calculated. Considering a 35% difference among groups to be significant, and a 95% probability of obtaining a significant difference among groups at the 5% level, the resulting number of subjects per group will be set 104.

To ensure an adequate quantity of surfaces at risk, participants will be required to have a minimum of 12 natural teeth.

Treatment The subjects will be randomly assigned to three groups: a Magnolia and Xylitol group (MX group) using a chewing gum containing MBE and xylitol, a Xylitol group (X group) using a chewing gum with the same content of xylitol but free of MBE and finally and a Control group (C group), using a sugar-free chewing gum without MBE and xylitol. Each subject will be instructed to chew 1 or 2 pellets for 5 minutes, 3 times a day (2 in the morning, 2 after the midday meal and 1 in the afternoon). Thus, the total daily intake of magnolol and honokiol in MX group will be 11.9 mg/day. The daily use of the three different chewing gums will be carried out for 12 months.

Three clinical evaluation for caries diagnosis will be performed: one at baseline, a second at the end of the chewing period (after 12 months from baseline) and a third after 24 months from baseline assessment. A microbiological evaluation for cariogenic bacteria will be performed immediately after the clinical assessments. Mutans streptococci and lactobacilli counts in saliva will be assessed and categorized using the dip-slide technique (CTR bacteria, Ivoclar Vivadent, Germany).

Following a sugar challenge, measures of interdental plaque pH, using pH indicator strips (Spezialindikator, pH range 4.0-7.0; Merck, Darmstadt, Germany), will be performed at 5 different points: at baseline, after 6 months of chewing gum use, after 12 months of chewing gum use, 6 months after the end of chewing gum use (18 months from baseline) and finally 12 months after the end of chewing gum use (24 months from baseline).

Randomization Eligible enrolees will be randomized to either the active or control arms. Randomization will be carried out using a computer-based program. Staff and participants will be blinded to treatment assignment.

Study Outcomes The primary study outcome will be the cumulative D2 or Filled Surface (D2 FS) increment (root and coronal surfaces combined) cumulated from baseline through the two follow-up examinations. In addition to the caries increment, data on participant safety and same risk factors related to caries development will be collected.

Expected results The results of this RCT should bring some clarity to the effectiveness of MBE as a caries preventive agent.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the recruitment of subjects are as follows:

1. Age 30-45
2. Presence of a minimum of 12 natural teeth
3. At least one surface cavitated caries lesion, but no more than three
4. Mutans streptococci and Lactobacilli >105 CFU/ml saliva
5. Systemically healthy as assessed by a medical questionnaire
6. No use of antibiotics or participation in a clinical study in the previous 30 days
7. No allergy to any of the ingredients of the study products
8. No orthodontic banding or removable prosthesis
9. Moderate gingivitis, no current periodontitis (no sites of probing pocket depth ≥5 mm or attachment loss of ≥2 mm, apart from gingival recession).
10. Absence of dysfunction of temporo-mandibular joint.

Exclusion Criteria:

* Subjects with a history of GI problems and with systemic disease that interfered with the oral ecosystem were excluded. The caries criterion was designed to include participants who are at risk of forming new lesions.
* In addition, those participants who were already consuming more than three pieces of sugar-free chewing gum a day were excluded.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
International Caries Detection and Assessment System (ICDAS) increment | 24 months
  cumulative D2 or Filled Surface (D2 FS) increment (root and coronal surfaces combined).

SECONDARY OUTCOMES:
Salivary mutants streptococci and lactobacilli counts | 6-12-24 months
  Mutans streptococci and lactobacilli counts in saliva were assessed
Modification of plaque pH | 6-12-24 months
  and categorized using the dip-slide technique Interproximal-plaque pH of each subject was evaluated using pH indicator strips, Assessment of plaque pH value in the range of 4.0-7.0.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Surgery, Microsurgery and Medicine Sciences University of Sassari, Sassari, Sardinia
  - WHO CC University of Milan, Milan

REFERENCES:
- [Derived] Cocco F, Carta G, Cagetti MG, Strohmenger L, Lingstrom P, Campus G. The caries preventive effect of 1-year use of low-dose xylitol chewing gum. A randomized placebo-controlled clinical trial in high-caries-risk adults. Clin Oral Investig. 2017 Dec;21(9):2733-2740. doi: 10.1007/s00784-017-2075-5. Epub 2017 Mar 16. PMID 28303470